CLINICAL TRIAL: NCT00888953
Title: Estudio de Medida Del Riesgo de Caídas Orientada a la Intervención en Residencias
Brief Title: Nursing Homes Study of Fall Risk Assessment Oriented to Intervention
Acronym: EMERCOIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Sociedad Española de Geriatría y Gerontología (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FICE09041; PI08/90162; 645H
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Accidental Falls; Activities of Daily Living; Quality of Life; Self-Efficacy
Keywords: Falls; Nursing Homes; Elderly; Prevention; Spain; Cluster Randomized Clinical Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Residents living in nursing homes allocated to intervention group. Assessment of risk factors. Implementation of a multifactorial tailored program to prevent falls.
  Interventions: Other: Fall risk assessment; Other: Tailored intervention
- Control (Other): Residents living in nursing homes allocated to control group. Assessment of risk factors. Receive the usual attention.
  Interventions: Other: Fall risk assessment

INTERVENTIONS:
Other: Fall risk assessment — Assessment of presence of risk factors (previous falls, self efficacy, balance and gait disorders, weakness, daily living impairment, limb pain, foot problems, dizziness, cognitive impairment, vision impairment, depression, urinary incontinence, heart disease, polimedication and consumption of neuroleptics and psychotropic medication)
  Other Names: Mini Falls Assessment (MFA)
Other: Tailored intervention — Induction of an intervention for each identified risk factor. If is possible the intervention will be directed towards the treatment of the underlying cause.
  Arms: Intervention

SUMMARY:
The aim of the study is to establish the impact of a falls screening questionnaire in the adoption of preventive interventions and eventually in the reduction of falls and its consequences in elder people living in nursing homes.

DETAILED DESCRIPTION:
Falls are the most frequent accidents in nursing homes, affecting more than a third of residents each year. Up to 10% of fallers require hospitalization or suffer a fracture. Psychological consequences affects between 20 and 80% of fallers, which suffer a lack of self-confidence that leads to reduction of activities and an increase of the dependence in activities of daily living.

Not all the residents have the same risk, and each person can have more than one risk factor that can be identified (previous falls, self confidence, weakness, gait disorders, dizziness, cognitive impairment, etc).

Identification of risk factors is the first step to reduce falls, but is not enough by itself. For this reason, interventions directed towards the correction of identified risk factors are required. In this setting, multifactorial interventions are the most successful to reduce falls numbers and its consequences.

As individual randomization of residents presents important inconveniences (group contamination, control arm residents could felt discriminated), we will randomized nursing homes to each group.

ELIGIBILITY:
Inclusion Criteria:

* People with or without cognitive impairment living indefinitely in a nursing home place
* Able to walk with or without any kind of help or able to self transfer (as defined in category d420 of the WHO International Classification of Functioning, Disability and Health) without help
* Give their consent (or the legal guardian in case of cognitive impairment).

Exclusion Criteria:

* Terminal illness (expected death before 6 months).
* Occupying temporarily a nursing home place (convalescence period) or another kind of place(day center, long term care, etc).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of fallers | one year
  People who at least have one fall during the follow-up period. Fall:unexpected event in which the participants come to rest on the ground, floor, or lower level

SECONDARY OUTCOMES:
Number of falls | one year
  Number of falls per person/time.
Number of people who has a fracture as a consequence of a fall | one year
Quality of life (only in residents without cognitive impairment). | One year
Activities of daily living | One year

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Salvà Casanovas, MD, Principal Investigator — Fundació Institut Català de l'Envelliment
Locations (1):
- Fundació Institut Català de l'Envelliment., Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Salva A, Rojano X, Coll-Planas L, Domenech S, Roque I Figuls M. [Randomized clinical trial of a fall-prevention strategy for institutionalized elderly based on the Mini Falls Assessment Instrument]. Rev Esp Geriatr Gerontol. 2016 Jan-Feb;51(1):18-24. doi: 10.1016/j.regg.2015.02.001. Epub 2015 Mar 14. Spanish. PMID 25777945